CLINICAL TRIAL: NCT07133282
Title: Functional Strength Building of Older Persons (FABULOS)
Brief Title: SingHealth Polyclinics - Functional Strength Building of Older Persons
Acronym: FABULOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SingHealth Polyclinics (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHPFABULOS
Record Dates: First submitted 2025-05-25; First posted 2025-08-21 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-04

CONDITIONS: Prefrail Elderly

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exercise group (Experimental): The intervention was twelve sessions of group exercise, delivered by exercise physiologists from ProAge (a health promotion social enterprise), lasting one hour each and conducted weekly. Each group had 10-15 participants. Nine sessions were held in-person, and three out of these twelve sessions were held remotely - the physiologist would send a video link of an exercise session for participants to follow at their own time for the week.
  Interventions: Behavioral: Group exercise programme

INTERVENTIONS:
Behavioral: Group exercise programme — 12-week group exercise programme

SUMMARY:
The goal of this study is to find out if a 12-week exercise programme for pre-frail seniors will result in an improvement in physical performance measures.

Participants attended 12 group exercise sessions, lasting one hour each, and held once a week. Three of these sessions were be conducted remotely, via a video link that participants will follow at their own time. Physical performance measures were taken at the first and last sessions.

ELIGIBILITY:
Inclusion Criteria:

* 65 years or older, and
* Clinical Frailty score of 3 or 4.

Exclusion Criteria:

* Persons who had pre-existing medical contraindications to exercise OR
* clinical symptoms that rendered them unsuitable for physical activity as determined by their attending physician OR
* cognitive impairment affecting their ability to provide informed consent.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 227 (Actual)
Dates: Start 2022-03-15 (Actual); Primary Completion 2023-06-08 (Actual); Study Completion 2024-01-16 (Actual)

PRIMARY OUTCOMES:
Short physical performance battery score | Assessed at baseline (at the start of the first exercise session) and 12 weeks (during the 12th exercise session)
  It assesses the functional mobility of an older adult's lower extremities in three domains (static balance, gait speed and chair stands). Balance is evaluated via the duration which participant can maintain side-by-side, semi-tandem, and tandem stances. Gait speed is measured by duration taken by the participant to walk 3 meters at their usual pace. Lower limb strength is assessed using the chair stand test, which records the time taken to complete five consecutive sit-to-stand movements from an armless chair with the participants' arms folded across the chest.
Hand grip strength | Assessed at baseline (at the start of the first exercise session) and 12 weeks (during the 12th exercise session)
  It is assessed using a handgrip dynamometer, with participants' elbows flexed at 90 degrees with the forearm in neutral position, squeezing the device as hard as possible with their left and right hands. The average recorded value from two measurements was used for analysis of this study
30-Seconds Sit-to-Stand repetitions | Assessed at first exercise session and 12th exercise session (i.e. 12 weeks from baseline)
  30-Seconds Sit-to-Stand repetitions is a measure of lower limb strength, endurance, and functional fitness. It is performed by recording the maximum number of times a participant can stand up fully and sit down from an armless chair within 30 seconds, with their arms folded across their chest. A higher number of repetitions indicate better functional capacity

SECONDARY OUTCOMES:
Change in exercise category in the International Physical Activity Questionnaire-Short Form (IPAQ-SF) | At enrolment, 6months post enrolment and 12 months post enrolment.
  Participants reported their physical activity based on an interviewer-administered IPAQ-SF during the enrolment visit, 6-month and 12-month after the start of the structured exercise programme.
  The IPAQ-SF is a validated instrument widely used as a measure of physical activity. The questionnaire contains 8 items, which assesses the frequency and duration of physical activity across domains such as sitting, walking, moderate-intensity activities and vigorous intensity activities. Based on the responses, the total metabolic equivalent (MET)-minutes per week is calculated, and participants are categorised into low, moderate, or high physical activity levels. There is no minimum or maximum value of MET-minutes per week as this is based on the participants' responses.

OTHER OUTCOMES:
Satisfaction scores | Administered at 12 weeks (i.e. at the 12th session).
  A researcher-developed satisfaction survey was used to assess participants' satisfaction with the sessions, instructors, venue, pace, exercises, and the perceived effects of FABULOS on their health.

CONTACTS AND LOCATIONS:
Overall Officials: Pei Lin Hu, MBBS, MMED(FM), FCFP(S), Principal Investigator — SingHealth Polyclinics
Locations (4):
- Singapore (4):
  - SingHealth Polyclinics - Marine Parade, Singapore, Singapore
  - SingHealth Polyclinics - Sengkang, Singapore, Singapore
  - SingHealth Polyclinics - Punggol, Singapore, Singapore
  - SingHealth Polyclinics - Tampines, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No
Sharing of IPD outside of the study team was not included in the informed consent form signed earlier by the participants.